CLINICAL TRIAL: NCT03306082
Title: Image-guided Cochlear Implant Programming (IGCIP)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jack Noble, Research Assistant Professor, Electrical Engineering and Computer Science, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150417; R01DC014037 (NIH)
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Intervention Model Description: Prospective Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Image-guided Cochlear Implant Programming (IGCIP) (Experimental): Cochlear implant programming using IGCIP.
  Interventions: Other: Image-Guided Cochlear Implant Programming

INTERVENTIONS:
Other: Image-Guided Cochlear Implant Programming — Post Cochlear Implant surgery, participant will receive traditional activation and programming per routine. IGCIP will be used to offer alternative programming of the implant.

SUMMARY:
Cochlear implants are surgically implanted devices which restore the ability to hear to the hearing impaired. While remarkably successful, even in the best of performers restoration of hearing to levels of normal listeners is unusual. Approximately 3 weeks after surgery, cochlear implants are activated via mapping - a process in which each individual electrode (FDA approved cochlear implants have between 12 and 22 electrodes) is turned on and the stimulus level adjusted to a level that is comfortable and beneficial to the recipient. At present, this standard of care mapping procedure is performed without knowledge of the physical location between the cochlear implant electrodes and the neural interface. The research team has developed a new method of mapping using post-operative CT scans and image processing to specify the physical relationship between the cochlear implant electrodes and the neural interface allowing customized mapping. Using this information, the investigators deactivate sub-optimally positioned electrodes. The investigators term this "Image-guided Cochlear Implant Programming" (IGCIP). The study collects data in a prospective fashion for those CI recipient undergoing IGCIP.

DETAILED DESCRIPTION:
Over 320,000 individuals have received cochlear implants (CIs) to restore hearing to the hearing impaired. Commercially available CIs have 12, 16, or 22 independent electrodes (the number is dependent on the manufacturer of the CI) which cover the entire frequency spectrum of the cochlea from 20,000 Hertz (Hz) at the base of to 200Hz at the apex. After implantation, an audiologist individually adjusts stimulation levels of each electrode following which all electrodes are turned on such that the whole frequency spectrum of speech can be appreciated. This is known as "standard of care" (SOC) programming. While postoperative speech understanding is significantly better than preoperative levels, even the best performers complain that the fidelity of natural hearing is not reproduced. Additionally, a significant minority achieves poor outcomes despite normally functioning equipment for reasons that are unknown but likely relate to poor neural survival; however, this cannot be confirmed as postmortem histopathology is required to accurately document spiral ganglion cell count. In recent years much attention has focused on the interface between the cochlear implant electrodes and the auditory neurons they are stimulating. Technological improvements at Vanderbilt in imaging processing have made it possible to determine the location of each electrode array in relationship to the frequency spectrum of the cochlea. Using this information, the investigators have developed a new method of CI programming which they call image-guided cochlear implant programming, or IGCIP in which sub-optimally placed electrodes are turned-off or deactivated. Sub-optimally placed electrodes are defined as ones for which their neighboring electrodes are in closer proximity to the site of their neural stimulation. By deactivating sub-optimally positioned electrodes, channel interaction is reduced allowing a cleaner signal to be presented to the auditory nerve. The purpose of the study is to prospectively collect audiological outcomes on patients undergoing IGCIP. The investigators hypothesize that CI recipients will perform better with IGCIP as compared to SOC.

Cochlear implant recipients who have reached asymptotic improvement in performance with SOC will be offered enrollment. They will undergo post-operative CT scanning to determine the relationship between the cochlear implant electrodes and the neural interface. Recommendations regarding deactivation of sub-optimally placed electrodes will be communicated to the audiology team who, if in their clinical judgement deems deactivation of these electrodes reasonable, will implement the changes for a 1 month trial. The participant will return at 1 month to have audiological assessment as per the clinical standard of care. Based on these results, which will be shared with the patient, the patient can choose to use IGCIP or SOC for long term cochlear implant programming.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 90 years that have undergone diagnostic testing for sensorineural hearing loss and have received a cochlear implant with asymptotic improvement in performance with SOC programming will be considered eligible for the study.

Exclusion Criteria:

* Age < 18 years or > 90 years
* Non-English speaking (because our audiological speech testing battery is validated for English speakers)
* Pregnancy which is a contraindication for elective CT scanning and surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-06-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
AzBio Sentence Scores at +5 Signal to Noise Ratio (SNR) | Month 1 post cochlear implant activation

SECONDARY OUTCOMES:
Minimum Speech Test Battery | Month 1 post cochlear implant activation

CONTACTS AND LOCATIONS:
Overall Officials: Jack H. Noble, PhD, Principal Investigator — Vanderbilt University; Rene H. Gifford, PhD, Study Chair — Vanderbilt University Medical Center; Robert F. Labadie, MD, PhD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No